CLINICAL TRIAL: NCT02540161
Title: Phase 2 Study of Sym004 for Adult Patients With Recurrent Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Annick Desjardins (Other)
Collaborators: Symphogen A/S (Industry)
Responsible Party: Sponsor-Investigator, Annick Desjardins, Associate Professor of Neurology, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00063483
Record Dates: First submitted 2015-09-01; First posted 2015-09-03 (Estimated); Results first posted 2020-07-24 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Malignant Glioma
Keywords: Sym004; Glioblastoma; Desjardins; Pro00063483; Symphogen; Duke Cancer Institute
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — futuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- non-bevacizumab failures - 18 mg/kg (Experimental): Non-bevacizumab failure (either no prior bevacizumab or bevacizumab stable/responder, which is defined as stable for at least 6 months from prior treatment with bevacizumab without experiencing a bevacizumab adverse event of special interest (AESI) while on a bevacizumab-containing regimen) will receive Sym004 intravenously every two weeks.
  Interventions: Drug: Sym004 - 18 mg/kg
- bevacizumab failures - 18 mg/kg (Experimental): Prior progression on a bevacizumab-containing regimen (defined as having progressed/grown through bevacizumab by RANO criteria within 2 months of prior bevacizumab treatment) will receive Sym004 intravenously every two weeks.
  Interventions: Drug: Sym004 - 18 mg/kg
- non-bevacizumab failures - 24 mg/kg (Experimental): Non-bevacizumab failure (either no prior bevacizumab or bevacizumab stable/responder, which is defined as stable for at least 6 months from prior treatment with bevacizumab without experiencing a bevacizumab adverse event of special interest (AESI) while on a bevacizumab-containing regimen) will receive Sym004 intravenously every two weeks.
  Interventions: Drug: Sym004 - 24 mg/kg
- bevacizumab failures - 24 mg/kg (Experimental): Prior progression on a bevacizumab-containing regimen (defined as having progressed/grown through bevacizumab by RANO criteria within 2 months of prior bevacizumab treatment) will receive Sym004 intravenously every two weeks.
  Interventions: Drug: Sym004 - 24 mg/kg

INTERVENTIONS:
Drug: Sym004 - 18 mg/kg — Sym004 was dosed at 18 mg/kg intravenously every two weeks.
  Arms: bevacizumab failures - 18 mg/kg; non-bevacizumab failures - 18 mg/kg
Drug: Sym004 - 24 mg/kg — Beginning in August 2017, the dose was increased to 24 mg/kg intravenously every two weeks.
  Arms: bevacizumab failures - 24 mg/kg; non-bevacizumab failures - 24 mg/kg

SUMMARY:
The purpose of this study is to assess the activity of Sym004, a recombinant antibody mixture that specifically binds to EGFR, in patients diagnosed with recurrent glioblastoma whose tumor is EGFR amplified. This is a phase 2 study that will accrue patients with WHO grade IV recurrent malignant glioma (glioblastoma or gliosarcoma) in two cohorts to assess the efficacy of Sym004.

DETAILED DESCRIPTION:
The purpose of this study is to assess the activity of Sym004, a recombinant antibody mixture that specifically binds to EGFR, in patients diagnosed with recurrent glioblastoma whose tumor is EGFR amplified. The primary objective is to assess the activity of Sym004 in patients with recurrent glioblastoma that are either non-bevacizumab failures (Cohort 1) or who have previously failed bevacizumab (Cohort 2), in terms of 6-month progression-free survival (PFS6). Secondary objectives include: 1. Determine the safety of Sym004 in recurrent glioblastoma (GBM) patients; 2. Estimate response rate (RR) within the two cohorts of recurrent GBM patients; 3. Describe overall survival (OS) within the two cohorts of recurrent GBM patients; 4. Describe overall median progress free survival (PFS) within the two cohorts of recurrent GBM patients.

This is a phase 2 study that will accrue patients with WHO grade IV recurrent malignant glioma (glioblastoma or gliosarcoma) in two cohorts to assess the efficacy of Sym004. Both cohorts will accrue simultaneously, with 36 subjects in Cohort 1 and 25 subjects in Cohort 2 at a dose of 18 mg/kg Sym004 given intravenously every 2 weeks. A treatment cycle will be 4 weeks.

Twenty-five subjects have been treated at the 18 mg/kg dose of Sym004. Beginning in August 2017, the dose of Sym004 will be increased to 24 mg/kg. Sixty-five additional subjects (36 in Cohort 1 and 29 in Cohort 2) will be treated at the new dose level.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed diagnosis of World Health Organization (WHO) grade 4 malignant glioma and radiographic evidence of recurrence or disease progression (as defined by the Response Assessment in Neuro-Oncology (RANO) criteria as a greater than 25% increase in the largest bi-dimensional product of enhancement or a new enhancing lesion, or a significant increase in T2-weighted-Fluid-Attenuated Inversion Recovery (T2/FLAIR) abnormality without another co-morbid cause);
2. Age ≥ 18 years;
3. Karnofsky Performance Status ≥ 70%;
4. No more than 3 prior progressions;
5. Cohort 1 only: Non-bevacizumab failure, i.e. either no prior bevacizumab or bevacizumab stable/responder, which is defined as stable within 6 months of prior treatment with bevacizumab without experiencing a bevacizumab adverse event of special interest (AESI) while on a bevacizumab-containing regimen, such as:

   1. ≥ grade 3 hypertension not controlled by medication, hypertensive crisis, or hypertensive encephalopathy
   2. ≥ grade 3 proteinuria that does not resolve or nephrotic syndrome
   3. Any grade GI perforation
   4. ≥ grade 3 infusion-related reaction
   5. ≥ grade 3 woundhealing complications
   6. ≥ grade 3 hemorrhage or any grade central nervous system (CNS) hemorrhage or ≥ grade 2 hemoptysis
   7. Any grade arterial thromboembolic event (e.g. myocardial infarction or cerebral infarction) or ≥ grade 3 venous thromboembolic event
   8. Any grade posterior reversible encephalopathy syndrome (PRES)
   9. ≥ grade 3 congestive heart failure
   10. ≥ grade 2 non-gastrointestinal (GI) abscesses and fistulae;
6. Cohort 2 only: Prior progression on a bevacizumab-containing regimen (defined as having progressed/grown through bevacizumab by RANO criteria within 2 months of prior bevacizumab treatment);
7. Pathology consistent with Epidermal Growth Factor Receptor (EGFR)-amplification of tumor (i.e. greater than 15% of cells exhibiting > 5 copies of EGFR loci); archival tissue may be tested for EGFR status in a separate consent;
8. Absolute Neutrophil Count (ANC) ≥ 1,000 cells/µl, platelets ≥ 100,000 cells/µl, hemoglobin ≥ 9 g/dL;
9. Adequate renal function as indicated by the following:

   1. Serum creatinine < 1.25 times upper limit of normal or calculated creatinine clearance ≥ 50 ml/min;
   2. Urine dipstick for proteinuria < 2+ unless a 24-hour urine protein <1 g of protein is demonstrated;
10. Adequate liver function as indicated by the following:

    1. Total bilirubin ≤ 1.6 mg/dL;
    2. Aspartate transaminase/alanine transaminase (AST/ALT) ≤ 2.5 x the upper limit of normal (ULN);
11. Magnesium ≥ 0.9 mg/dL;
12. For subjects on corticosteroids, they must be on a stable dose for 7 days prior to anticipated start of study drug;
13. No evidence of > grade 1 active CNS hemorrhage on the baseline magnetic resonance imaging (MRI) or X-ray computed tomography (CT) scan;
14. Signed informed consent approved by the Institutional Review Board prior to patient entry;
15. If the patient is a sexually active female of child bearing potential whose partner is male, or if the patient is a sexually active male whose partner is a female of child bearing potential, the patient must agree to use appropriate contraceptive measures for the duration of the treatment of the tumor and for 6 months afterwards as stated in the informed consent. Female patients of child bearing potential must have a negative serum pregnancy test within 48 hours of starting study treatment;
16. Fertile male subjects must agree to use a medically acceptable contraceptive method (allowed methods of birth control include vasectomy or condom with spermicide) during the trial and for a period of at least 6 months following the last administration of trial drugs.

Exclusion Criteria:

1. Pregnancy or breastfeeding;
2. Prior treatment with EGFR-targeted therapy, including, but not limited to, the following examples: Gilotrif® (afatinib),Tarceva® (erlotinib), Erbitux® (cetuximab), Iressa™ (gefitinib), Vectibix® (panitumumab), Caprelsa® (vandetanib), Tykerb® (lapatinib), CDX110, D2C7-immunotoxin;
3. Active infection requiring intravenous antibiotics within 7 days before enrollment;
4. Prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin;
5. Less than 12 weeks from radiation therapy, unless progressive disease outside of the radiation field or 2 progressive scans at least 4 weeks apart or histopathologic confirmation;
6. Treated with immunotherapeutic agents, vaccines, or Mab therapy within 4 weeks before enrollment, unless the patient has recovered from the expected toxic effects of such therapy
7. Treated with alkylating agents within 4 weeks (6 weeks for nitrosoureas) before enrollment or treated within 1 week before enrollment with daily or metronomic chemotherapy, unless the patient has recovered from the expected toxic effects of such therapy to their baseline or to grade 1;
8. Prior treatment (non-alkylating agents) within 2 weeks before enrollment, unless the patient has recovered from the expected toxic effects of such therapy;
9. Known hypersensitivity reactions to any of the components of Sym004;
10. Known current drug abuse or alcohol abuse;
11. Known Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C infection. Testing is not required as part of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2020-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annick Desjardins, MD, FRCPC, Principal Investigator — Duke University
Locations (1):
- The Preston Robert Tisch Brain Tumor Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at Duke — https://tischbraintumorcenter.duke.edu/
- See also: Duke Cancer Institute — http://www.dukecancerinstitute.org/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 43 patients signed consent and were considered enrolled, however 3 patients withdrew consent prior to treatment and 1 patient was withdrawn by PI prior to treatment.
Period: Overall Study
Arm/Group | Non-bevacizumab Failures - 18 mg/kg | Bevacizumab Failures - 18 mg/kg | Non-bevacizumab Failures - 24 mg/kg | Bevacizumab Failures - 24 mg/kg
Started | 20 | 7 | 5 | 7
Completed | 20 | 7 | 5 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-bevacizumab Failures - 18 mg/kg | Bevacizumab Failures - 18 mg/kg | Non-bevacizumab Failures - 24 mg/kg | Bevacizumab Failures - 24 mg/kg | Total
Number analyzed (Participants) | 20 | 7 | 5 | 7 | 39
Age, Continuous [Median (Full Range); unit: years] | 58.5 [34 to 72] | 53 [41 to 76] | 61 [39 to 71] | 56 [51 to 72] | 57.25 [34 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 0 | 2 | 15
  Male | 10 | 4 | 5 | 5 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 6 | 5 | 7 | 38
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 19 | 7 | 4 | 7 | 37
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 7 | 5 | 7 | 39

OUTCOME MEASURES:

1. Primary Outcome: Six-month Progression-free Survival (PFS6)
Description: Within each cohort, the percentage of participants alive and progression-free at 6 months after the start of Sym004 treatment will be determined. PFS6 will be calculated from the date study treatment started until the date of progression or death, or the date of last follow-up if participants are alive without progression. Kaplan-Meier methods will be used to estimate survival.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Non-bevacizumab Failures - 18 mg/kg | Bevacizumab Failures - 18 mg/kg | Non-bevacizumab Failures - 24 mg/kg | Bevacizumab Failures - 24 mg/kg
Number analyzed (Participants) | 20 | 7 | 5 | 7
percentage of participants | 14.3 [0.7 to 46.5] | 5 [0.3 to 20.5] | 14.3 [0.7 to 46.5] | 40 [5.2 to 75.3]

2. Secondary Outcome: Percentage of Participants Who Experience Grade 3, 4 or 5 Adverse Events
Description: Within each cohort, the percentage of participants who experience grade 3, 4 or 5 adverse events that are possibly, probably or definitely related to study treatment will be calculated.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Non-bevacizumab Failures - 18 mg/kg | Bevacizumab Failures - 18 mg/kg | Non-bevacizumab Failures - 24 mg/kg | Bevacizumab Failures - 24 mg/kg
Number analyzed (Participants) | 20 | 7 | 5 | 7
percentage of participants | 15 | 42.86 | 40 | 14.29

3. Secondary Outcome: Radiographic Response
Description: Within each cohort, the percentage of participants with a complete or partial response as determined by modified Response Assessment in Neuro-Oncology (RANO) criteria will be determined. Complete Response (CR) is defined as complete disappearance on MR/CT of all enhancing tumor and mass effect, off all corticosteroids (or receiving only adrenal replacement doses) and accompanied by a stable or improving neurologic examination. Partial Response (PR) is defined as greater than or equal to 50% reduction in tumor size on MR/CT by bi-dimensional measurement, on a stable or decreasing dose of corticosteroids and accompanied by a stable or improving neurologic examination. Tumor assessments are done at baseline and the end of every second cycle (every 8 weeks) thereafter.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Non-bevacizumab Failures - 18 mg/kg | Bevacizumab Failures - 18 mg/kg | Non-bevacizumab Failures - 24 mg/kg | Bevacizumab Failures - 24 mg/kg
Number analyzed (Participants) | 20 | 7 | 5 | 7
percentage of participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Median Progression-free Survival (PFS)
Description: Median PFS will be estimated within each cohort. Progression-free survival is defined as the time in months from the start of protocol treatment until the date of progression or death if death occurred before progression. If the participant is alive and progression-free, PFS will be censored at the date of last follow-up. Kaplan-Meier methods will be used to estimate progression-free survival.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Non-bevacizumab Failures - 18 mg/kg | Bevacizumab Failures - 18 mg/kg | Non-bevacizumab Failures - 24 mg/kg | Bevacizumab Failures - 24 mg/kg
Number analyzed (Participants) | 20 | 7 | 5 | 7
months | 1.81 [1.35 to 2.43] | 3.91 [1.51 to 5.79] | 3.55 [0.65 to 11.27] | 2.00 [0.85 to 2.20]

5. Secondary Outcome: Median Overall Survival (OS)
Description: Median OS will be estimated within each cohort. Overall survival is defined as the time in months from the start of protocol treatment until the date of death, or the date of last follow-up if alive. Kaplan-Meier methods will be used to estimate overall survival.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Non-bevacizumab Failures - 18 mg/kg | Bevacizumab Failures - 18 mg/kg | Non-bevacizumab Failures - 24 mg/kg | Bevacizumab Failures - 24 mg/kg
Number analyzed (Participants) | 20 | 7 | 5 | 7
months | 7.54 [3.88 to 10.81] | 5.51 [1.87 to 8.80] | 9.95 [4.17 to 15.54] | 5.39 [0.85 to 8.64]

ADVERSE EVENTS:
Time Frame: From the start of study treatment for a patient until 30 days after treatment is discontinued, maximum of 1 year.
Description: Patients were evaluated for adverse events (all grades), serious adverse events, and adverse events requiring study drug interruption or discontinuation at each study visit for the duration of their participation in the study.
Groups:
- Non-bevacizumab Failures - 18 mg/kg: Non-bevacizumab failure (either no prior bevacizumab or bevacizumab stable/responder, which is defined as stable for at least 6 months from prior treatment with bevacizumab without experiencing a bevacizumab adverse event of special interest (AESI) while on a bevacizumab-containing regimen) will receive Sym004 intravenously every two weeks.
  Sym004: Sym004 was dosed at 18 mg/kg intravenously every two weeks.
- Bevacizumab Failures - 18 mg/kg: Prior progression on a bevacizumab-containing regimen (defined as having progressed/grown through bevacizumab by RANO criteria within 2 months of prior bevacizumab treatment) will receive Sym004 intravenously every two weeks.
  Sym004: Sym004 was dosed at 18 mg/kg intravenously every two weeks. .
- Non-bevacizumab Failures - 24 mg/kg: Non-bevacizumab failure (either no prior bevacizumab or bevacizumab stable/responder, which is defined as stable for at least 6 months from prior treatment with bevacizumab without experiencing a bevacizumab adverse event of special interest (AESI) while on a bevacizumab-containing regimen) will receive Sym004 intravenously every two weeks.
  Beginning in August 2017, the dose was increased to 24 mg/kg intravenously every two weeks.
- Bevacizumab Failures - 24 mg/kg: Prior progression on a bevacizumab-containing regimen (defined as having progressed/grown through bevacizumab by RANO criteria within 2 months of prior bevacizumab treatment) will receive Sym004 intravenously every two weeks.
  Beginning in August 2017, the dose was increased to 24 mg/kg intravenously every two weeks.
Arm/Group | Non-bevacizumab Failures - 18 mg/kg | Bevacizumab Failures - 18 mg/kg | Non-bevacizumab Failures - 24 mg/kg | Bevacizumab Failures - 24 mg/kg
All-Cause Mortality (participants affected / at risk) | 20/20 | 7/7 | 5/5 | 7/7
Serious Adverse Events (participants affected / at risk) | 8/20 | 2/7 | 2/5 | 4/7
Other Adverse Events (participants affected / at risk) | 20/20 | 7/7 | 5/5 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-bevacizumab Failures - 18 mg/kg (N=20) | Bevacizumab Failures - 18 mg/kg (N=7) | Non-bevacizumab Failures - 24 mg/kg (N=5) | Bevacizumab Failures - 24 mg/kg (N=7)
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Edema limbs (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 0
Catheter related infection (Infections and infestations) | 1 | 0 | 0 | 0
Infections and infestations - Other, Specify: FEVER (Infections and infestations) | 0 | 1 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 1 | 0 | 0
Papulopustular rash (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Injury, poisoning and procedural complications - Other, Specify: CHARGED/HEADBUTTED BY BULL (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 — "FACE SWOLLEN", "BLOODY AND RAW", "SLOUGHING OFF"
Dysphasia (Nervous system disorders) | 1 | 1 | 0 | 0
Seizure (Nervous system disorders) | 4 | 0 | 2 | 1
Confusion (Psychiatric disorders) | 1 | 0 | 0 | 0
Renal and urinary disorders - Other, Specify: NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-bevacizumab Failures - 18 mg/kg (N=20) | Bevacizumab Failures - 18 mg/kg (N=7) | Non-bevacizumab Failures - 24 mg/kg (N=5) | Bevacizumab Failures - 24 mg/kg (N=7)
Anemia (Blood and lymphatic system disorders) | 3 | 1 | 2 | 1
Cardiac disorders - Other, Specify: TACHYCARDIA (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Ear and labyrinth disorders - Other, Specify: "EAR FULLNESS/SWELLING" FEELING (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Ear and labyrinth disorders - Other, Specify: EAR DISCHARGE (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Ear and labyrinth disorders - Other, Specify: INTERMITTENT FEELING OF WATER IN EARS (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Blurred vision (Eye disorders) | 1 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 1 | 1 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0
Eye disorders - Other, Specify: "BLURRED", EYES CLOSED MOST TIMES (Eye disorders) | 0 | 0 | 0 | 1
Eye disorders - Other, Specify: DECREASED VISION (Eye disorders) | 1 | 0 | 0 | 0
Eye disorders - Other, Specify: DIPLOPIA (Eye disorders) | 0 | 0 | 1 | 0
Eye disorders - Other, Specify: EYELID ITCHING, RIGHT EYE REDNESS, CRUSTING TO EYES (Eye disorders) | 0 | 0 | 1 | 0
Eye disorders - Other, Specify: HEMIANOPIA (Eye disorders) | 0 | 0 | 1 | 0
Eye disorders - Other, Specify: L EYE WITH DRAINAGE; CRUST AROUND EYELID (Eye disorders) | 0 | 1 | 0 | 0
Anal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 1 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Fecal incontinence (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal disorders - Other, Specify: GLOSSITIS (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal disorders - Other, Specify: HYPERSALIVATION (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal disorders - Other, Specify: MOUTH SORES (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 0 | 1 | 1
Oral hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 2 | 0
Edema face (General disorders) | 1 | 0 | 1 | 0
Edema limbs (General disorders) | 1 | 0 | 0 | 1
Fatigue (General disorders) | 7 | 2 | 3 | 2
Flu like symptoms (General disorders) | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 1 | 1 | 1 | 0
General disorders and administration site conditions - Other, Specify: CHILLS (General disorders) | 0 | 0 | 1 | 0
General disorders and administration site conditions - Other, Specify: RUNNY NOSE (General disorders) | 0 | 0 | 1 | 0
Infusion related reaction (General disorders) | 3 | 2 | 1 | 2
Irritability (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 4 | 0 | 2 | 2
Infections and infestations - Other, Specify: BACTEREMIA (Infections and infestations) | 1 | 0 | 0 | 0
Infections and infestations - Other, Specify: FUNGAL RASH (Infections and infestations) | 1 | 0 | 0 | 0
Infections and infestations - Other, Specify: MRSA INFECTION (Infections and infestations) | 0 | 0 | 1 | 0
Mucosal infection (Infections and infestations) | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0
Papulopustular rash (Infections and infestations) | 2 | 1 | 0 | 1
Paronychia (Infections and infestations) | 0 | 1 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 3 | 1 | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 0
Burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 0 | 1 | 1
Injury, poisoning and procedural complications - Other, Specify: LACERATION TO RIGHT LOWER LEG (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Injury, poisoning and procedural complications - Other, Specify: WOUND FROM FALL; DRAINAGE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 2 | 0 | 2
Alkaline phosphatase increased (Investigations) | 4 | 2 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1 | 2
Creatinine increased (Investigations) | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 5 | 1 | 1 | 2
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 2
Platelet count decreased (Investigations) | 1 | 1 | 0 | 4
Weight loss (Investigations) | 0 | 1 | 0 | 0
White blood cell decreased (Investigations) | 1 | 1 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 8 | 2 | 4 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 | 3 | 3 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 8 | 3 | 4 | 4
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 8 | 2 | 1 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 13 | 5 | 4 | 3
Hyponatremia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 2
Dysphasia (Nervous system disorders) | 3 | 1 | 0 | 1
Headache (Nervous system disorders) | 7 | 2 | 2 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 1 | 2
Nervous system disorders - Other, Specify: DIFFICULTY HOLDING ITEMS WITH HIS LEFT HAND (Nervous system disorders) | 0 | 0 | 1 | 0
Nervous system disorders - Other, Specify: DISORIENTATION (Nervous system disorders) | 0 | 0 | 1 | 0
Nervous system disorders - Other, Specify: WEAKNESS, BALANCE OFF (Nervous system disorders) | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 2
Pyramidal tract syndrome (Nervous system disorders) | 1 | 0 | 1 | 1
Seizure (Nervous system disorders) | 6 | 4 | 2 | 1
Tremor (Nervous system disorders) | 0 | 1 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Confusion (Psychiatric disorders) | 1 | 0 | 1 | 3
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Hematuria (Renal and urinary disorders) | 2 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 2 | 1 | 0
Renal and urinary disorders - Other, Specify: DISCOLORED URINE (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 1 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 1 | 1 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 4 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 | 0 | 2 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 | 6 | 4 | 4
Skin and subcutaneous tissue disorders - Other, Specify: INDEX FINGER CUTICLE REDNESS/IRRITATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, Specify: "BRUISING APPEARANCE" (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin and subcutaneous tissue disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 — "FACE SWOLLEN", "BLOODY AND RAW", "ALMOST SLOUGHING OFF"
Skin and subcutaneous tissue disorders - Other, Specify: "REDNESS TO CHEEKS" (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 — "RIGHT HAND NEAR NAIL BEDS", "CRUSTING", "PAINFUL/BURNING"
Skin and subcutaneous tissue disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 — BLEEDING FROM CRACKS ON EARS, "STAINING LARGE AREAS OF PILLOWCASES"
Skin and subcutaneous tissue disorders - Other, Specify: FACIAL REDNESS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 — FINGERNAIL BEDS AND TIPS OF FINGERS CRACKING AND PAINFUL TO TOUCH
Skin and subcutaneous tissue disorders - Other, Specify: HEELS CRACKED WITH SCABBING AND BRUISING (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 — PEELING SKIN, FACIAL AREA ALONG EYES, NOSE, AND MOUTH AREA
Skin and subcutaneous tissue disorders - Other, Specify: RASH (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 0
Skin and subcutaneous tissue disorders - Other, Specify: RED PATCHY SPOTS/WHITE HEAD ON NOSE (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, Specify: SENSITIVE FEET (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, Specify: SKIN TEARS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, Specify: SKIN TRAUMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, Specify: SOME NAILBEDS OF FINGERS REDDENED (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin and subcutaneous tissue disorders - Other, Specify: SORE, INFLAMED AREA BEHIND L EAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, Specify: SUNBURN (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT02540161/Prot_SAP_000.pdf